CLINICAL TRIAL: NCT01744457
Title: Reproducibility of Tearfilm Osmolarity Measurements Using TearLab® in Patients With Dry Eye Syndrome and Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OPHT-161009
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Dry Eye Syndrome
Keywords: tear film osmolarity; objective scattering index; tear break up time; Schirmer I test
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 20 patients with dry eye syndrome (Other): Patients with dry eye syndrome defined as outlined in the inclusion and exclusion criteria
  Interventions: Device: Measurement of tear film osmolarity with the TearLab® instrument; Other: Schirmer I test; Other: Tear break up time; Device: Optical Quality Analysis System; Other: Ocular Surface Disease Index
- 20 healthy control subjects (Other): age- and sex-matched controls
  Interventions: Device: Measurement of tear film osmolarity with the TearLab® instrument; Other: Schirmer I test; Other: Tear break up time; Device: Optical Quality Analysis System; Other: Ocular Surface Disease Index

INTERVENTIONS:
Device: Measurement of tear film osmolarity with the TearLab® instrument
Other: Schirmer I test
Other: Tear break up time
Device: Optical Quality Analysis System — Measurement of the objective scattering index (OSI)
Other: Ocular Surface Disease Index

SUMMARY:
Dry Eye Syndrome (DES) is a common condition that affects approximately 20% of adults aged 45 and older. Although several clinical tests for the diagnosis and monitoring of DES are available, currently no gold standard for the assessment of DES exists. It has, however, been hypothesized that the assessment of tear film osmolarity may be a new and promising approach of an objective and non-invasive method for diagnosis and monitoring of treatment success.

Recently, a new commercially available instrument (TearLab®, OcuSens Inc, San Diego, USA) for the assessment of tear film osmolarity has been introduced. This instrument allows for the easy and non-invasive determination of tear film osmolarity. Unfortunately, no data about reproducibility are yet available. Consequently, the current study sets out to investigate the short time reproducibility of tear film osmolarity measurements using the TearLab® instrument.

ELIGIBILITY:
Inclusion Criteria:

Patients with dry eye syndrome (DES):

* Men and Women aged between 45 and 80 years, with DES defined as a pathological Schirmer I test and / or a pathological break-up time test. Schirmer I test and break up time will be tested and analyzed according to the guidelines published in the Report of the International Dry EyeWorkShop (DEWS) 2007
* normal findings in the ophthalmic examination other than DES

Healthy control group:

* Men and Women aged between 45 and 80 years,
* normal findings in the medical history and ophthalmic examination

Exclusion Criteria:

* Abuse of drugs or alcoholic beverages
* Participation in a clinical trial
* Symptoms of a clinically relevant illness

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Coefficient of variation of tear film osmolarity after repeated measurements | Measurement of tear film osmolarity 3 times daily within 30 minutes for 3 consecutive days

SECONDARY OUTCOMES:
Subjective symptoms assessed using the OSDI test | on the screening day
Tear break up time | on 3 consecutive study days once a day
Schirmer I test | on 3 consecutive study days once a day
OSI (Objective Scattering Index) | on 3 consecutive study days once a day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria